CLINICAL TRIAL: NCT02686021
Title: Potential Benefit of the Combination of Metamizole and Ibuprofen After Third Lower Molar Extraction
Acronym: NovIbu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKNZ 2015-284
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dipyrone; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metamizole and Ibuprofen (Experimental): all patients (n=42) will receive metamizol and ibuprofen in one session. In the other session half will receive metamizol and placebo (n=21) and the other half will receive ibuprofen and placebo. The order will be randomized (balanced).
  Interventions: Drug: Metamizole and Ibuprofen
- Metamizole and Placebo (Active Comparator): This is one of the two comparators for the Arm "Metamizol and Ibuprofen". n=21
  Interventions: Drug: Metamizole and Placebo
- Ibuprofen and Placebo (Active Comparator): This is the second of the two comparators for the Arm "Metamizol and Ibuprofen". n=21
  Interventions: Drug: Ibuprofen and Placebo

INTERVENTIONS:
Drug: Metamizole and Ibuprofen — Metamizole (1000mg) plus Ibuprofen (400mg) 15 minutes prior to surgery, at 6 postoperative hours, and at 12 postoperative hours
  Arms: Metamizole and Ibuprofen
Drug: Metamizole and Placebo — Metamizole (1000mg) plus placebo 15 minutes prior to surgery, at 6 postoperative hours, and at 12 postoperative hours
  Arms: Metamizole and Placebo
Drug: Ibuprofen and Placebo — Ibuprofen (400mg) plus placebo 15 minutes prior to surgery, at 6 postoperative hours, and at 12 postoperative hours
  Arms: Ibuprofen and Placebo

SUMMARY:
Postoperative pain is common and particularly outpatients may experience unsatisfactory pain relief. This randomized, double-blind, crossover study of postoperative pain in outpatients undergoing split-mouth, third lower molar extraction aims to examine whether or not the combination of metamizole and ibuprofen is superior to either drug alone.

ELIGIBILITY:
Inclusion Criteria:

* planned sequential both-sided lower third molar extraction (split-mouth) with osteotomy (with or without upper molar extraction in local anesthesia)
* able to understand the study and the NRS scale

Exclusion Criteria:

* simultaneous both sided extraction or only upper third molar extraction
* general anesthesia
* known or presumed abnormal coagulation status
* known or presumed liver or renal dysfunction
* contraindication against metamizole known or suspected (known or suspected allergy against novalgin or other pyrazolones, anaphylactic reaction against NSAIDS, decreased bone marrow function or hematopoesis, hepatic porphyria, glucose-6-phosphate dehydrogenase deficiency, and pregnancy/breastfeeding)
* contraindication against ibuprofen (known or suspected allergy against ibuprofen, anaphylactic reaction against Nonsteroidal anti-inflammatory drugs (NSAID), active or recurrent stomach or duodenal ulcera or bleeding, severe liver or renal insufficiency, inflammatory bowel syndrome, and pregnancy/breastfeeding)
* pregnancy and breast feeding mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
area under the curve for pain in the first 12 postoperative hours | first 12 postoperative hours
  The primary outcome is the area under the curve for pain in the first 12 postoperative hours, as assessed by the numeric rating scale

SECONDARY OUTCOMES:
area under the curve for pain in the first 18 postoperative hours | first 18 postoperative hours
  This secondary outcome is the area under the curve for pain in the first 18 postoperative hours, as assessed by the numeric rating scale (NRS)
highest pain score | total observation period (maximum 18 hours)
  This secondary outcome is the highest pain score registered during the observation period, as assessed by the numeric rating scale
night time pain | first night after the intervention
  This secondary outcome is the overall pain during the first night after the intervention, as assessed by the numeric rating scale
need for and timing of rescue medication | total observation period (maximum 18 hours)
  This secondary outcome is the marked "yes" or "no", depending on whether a rescue medication (extra pain medication) was needed or not
haemorrhage requiring intervention | total observation period (maximum 18 hours)
  This secondary outcome is the marked "yes" or "no", depending on whether an intervention to stop haemorrhage was needed or not

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Anesthesia, University of Basel Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided